CLINICAL TRIAL: NCT07178548
Title: Assessing Compliance With Low Back Pain Treatment Guidelines: Attitudes of Physiotherapists and Internship Students
Brief Title: Understanding How Physiotherapists in Türkiye Follow Low Back Pain Guidelines and What Affects Their Use of Research in Practice
Status: Enrolling by invitation | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Talat Abdelfatah Elnabawy, Principal Investigator, Medipol University
Other Study IDs: E-10840098-202.3.02-3367
Record Dates: First submitted 2025-06-29; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Guideline Adherence; Physiotherapist; Physiotherapist Students
Keywords: Low back pain; LBP; Physiotherapy; Physical therapy; Evidence-Based Practice; Türkiye; Physiotherapy Interns; Survey Study; Guideline Adherence
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Licenced Physiotherapists: This group includes licenced physical therapists currently practicing in Turkey in various settings, such as hospitals, private clinics rehabilitation centers or universities.
  Interventions: Other: Online Survey
- Intern Physiotherapists: This group includes physiotherapy students in their clinical internship period from accredited universities in Turkey.
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Participants will complete a structured online survey designed to assess their knowledge, attitudes, and application of evidence-based guidelines (clinical practice guidelines - CPGs) in managing low back pain (LBP).

SUMMARY:
The goal of this observational study is to understand how physiotherapists and physiotherapy students in Türkiye manage low back pain and how closely they follow clinical practice guidelines and use research evidence.

The main questions it aims to answer are:

* Do physiotherapists follow evidence-based guidelines when treating low back pain?
* What factors influence their treatment choices and use of research in practice?

Participants will:

* Complete a short online survey (about 5-10 minutes)
* Answer questions about their education, clinical decisions, and treatment approaches for low back pain

ELIGIBILITY:
Inclusion Criteria:

* Be a licensed physiotherapist currently practicing in Türkiye OR be a physiotherapy intern student enrolled in a clinical internship in Türkiye
* Have experience managing patients with low back pain (LBP)
* Ability to provide informed consent and complete an online questionnaire.

Exclusion Criteria:

* Are not currently practicing physiotherapy or not currently enrolled in a clinical internship
* Have no experience in managing low back pain patients
* Are unable to complete an online questionnaire due to technological or literacy limitations
* Decline to provide informed consen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from hospitals, rehabilitation centers, private clinics, and university physiotherapy programs across Türkiye. The population includes licensed physiotherapists and final-year physiotherapy students involved in low back pain rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Level of Adherence to Clinical Practice Guidelines (CPGs) for Low Back Pain (LBP) Rehabilitation | At the time of survey completion (Baseline)
  Assessment of the level of adherence to evidence-based LBP rehabilitation guidelines among licensed physical therapists and 4th-year internship students. This is measured by responses to a structured questionnaire evaluating compliance with specific clinical practice recommendations.
Comparison of Guideline Adherence Between Licensed Physical Therapists and Internship Students | At the time of survey completion (baseline)
  Analysis of differences in adherence scores between licensed physical therapists and internship students to identify any significant variation in the implementation of guideline practices.

SECONDARY OUTCOMES:
Perceived Barriers to Implementing Evidence-Based Practice (EBP) | At the time of survey completion (Baseline)
  Evaluation of the challenges and barriers reported by physical therapists and internship students in applying evidence-based stroke rehabilitation guidelines and advanced techniques, as gathered through the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, Dr. Assistant Professor, Study Director — Department of Physiotherapy and Rehabilitation/Istanbul Medipol University
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aytar, A., Çağlar, A., Tekindal, M. A., Ümit Yemişçi, O., et al. (2023). EFFECTIVENESS OF DIFFERENT PHYSICAL THERAPY EXERCISE TECHNIQUES IN CHRONIC LOW BACK PAIN: A RANDOMIZED CONTROLLED STUDY. Türk Fizyoterapi Ve Rehabilitasyon Dergisi, 34(1), 141-147. https://doi.org/10.21653/tjpr.1034741
- [Background] Anar SO. The effectiveness of home-based exercise programs for low back pain patients. J Phys Ther Sci. 2016 Oct;28(10):2727-2730. doi: 10.1589/jpts.28.2727. Epub 2016 Oct 28. PMID 27821923
- [Background] Schuster S, Loncaric Kelecic I, Bilic M, Begic M, Pate JW. Conceptualization of pain in Croatian adults: a cross-sectional and psychometric study. Croat Med J. 2024 Dec 30;65(6):473-482. doi: 10.3325/cmj.2024.65.472. PMID 39812096
- [Background] Scott NA, Moga C, Harstall C. Managing low back pain in the primary care setting: the know-do gap. Pain Res Manag. 2010 Nov-Dec;15(6):392-400. doi: 10.1155/2010/252695. PMID 21165374
- [Background] Rutten GM, Degen S, Hendriks EJ, Braspenning JC, Harting J, Oostendorp RA. Adherence to clinical practice guidelines for low back pain in physical therapy: do patients benefit? Phys Ther. 2010 Aug;90(8):1111-22. doi: 10.2522/ptj.20090173. Epub 2010 May 20. PMID 20488978
- [Background] Custers P, Van de Kelft E, Eeckhaut B, Sabbe W, Hofman A, Debuysscher A, Van Acker G, Maes G. Clinical Examination, Diagnosis, and Conservative Treatment of Chronic Low Back Pain: A Narrative Review. Life (Basel). 2024 Aug 29;14(9):1090. doi: 10.3390/life14091090. PMID 39337874
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Guzman J, Esmail R, Karjalainen K, Malmivaara A, Irvin E, Bombardier C. Multidisciplinary rehabilitation for chronic low back pain: systematic review. BMJ. 2001 Jun 23;322(7301):1511-6. doi: 10.1136/bmj.322.7301.1511. PMID 11420271
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain. Cochrane Database Syst Rev. 2014 Sep 2;2014(9):CD000963. doi: 10.1002/14651858.CD000963.pub3. PMID 25180773
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Pincus T, Kent P, Bronfort G, Loisel P, Pransky G, Hartvigsen J. Twenty-five years with the biopsychosocial model of low back pain-is it time to celebrate? A report from the twelfth international forum for primary care research on low back pain. Spine (Phila Pa 1976). 2013 Nov 15;38(24):2118-23. doi: 10.1097/BRS.0b013e3182a8c5d6. PMID 23970112
- [Background] Shiri R, Karppinen J, Leino-Arjas P, Solovieva S, Viikari-Juntura E. The association between smoking and low back pain: a meta-analysis. Am J Med. 2010 Jan;123(1):87.e7-35. doi: 10.1016/j.amjmed.2009.05.028. PMID 20102998
- [Background] Karahan A, Kav S, Abbasoglu A, Dogan N. Low back pain: prevalence and associated risk factors among hospital staff. J Adv Nurs. 2009 Mar;65(3):516-24. doi: 10.1111/j.1365-2648.2008.04905.x. PMID 19222649
- [Background] Celik S, Celik K, Dirimese E, Tasdemir N, Arik T, Buyukkara I. Determination of pain in musculoskeletal system reported by office workers and the pain risk factors. Int J Occup Med Environ Health. 2018 Jan 1;31(1):91-111. doi: 10.13075/ijomeh.1896.00901. Epub 2017 Oct 2. PMID 28972599
- [Background] Capkin E, Karkucak M, Cakirbay H, Topbas M, Karaca A, Kose MM, Gokmen F. The prevalence and risk factors of low back pain in the eastern Black Sea region of Turkey. J Back Musculoskelet Rehabil. 2015;28(4):783-7. doi: 10.3233/BMR-150584. PMID 25736952
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Transl Med. 2020 Mar;8(6):299. doi: 10.21037/atm.2020.02.175. PMID 32355743
- [Background] Koes BW, van Tulder M, Lin CW, Macedo LG, McAuley J, Maher C. An updated overview of clinical guidelines for the management of non-specific low back pain in primary care. Eur Spine J. 2010 Dec;19(12):2075-94. doi: 10.1007/s00586-010-1502-y. Epub 2010 Jul 3. PMID 20602122
- [Background] Dionne CE, Dunn KM, Croft PR, Nachemson AL, Buchbinder R, Walker BF, Wyatt M, Cassidy JD, Rossignol M, Leboeuf-Yde C, Hartvigsen J, Leino-Arjas P, Latza U, Reis S, Gil Del Real MT, Kovacs FM, Oberg B, Cedraschi C, Bouter LM, Koes BW, Picavet HS, van Tulder MW, Burton K, Foster NE, Macfarlane GJ, Thomas E, Underwood M, Waddell G, Shekelle P, Volinn E, Von Korff M. A consensus approach toward the standardization of back pain definitions for use in prevalence studies. Spine (Phila Pa 1976). 2008 Jan 1;33(1):95-103. doi: 10.1097/BRS.0b013e31815e7f94. PMID 18165754